CLINICAL TRIAL: NCT05412251
Title: Smart Integrated Health Promotion Program and Health Behavior for Older Adult
Brief Title: Smart Integrated Health Promotion Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YM110168-EF
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-02

CONDITIONS: Quality of Life
Keywords: leisure activity; nutrition status; quality of life; subjective well-being; older adults

STUDY DESIGN:
Intervention Model Description: control group and experimental group
Who Masked: Participant
Masking Description: control group and experimental group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- contrl (No Intervention): provide an irregular nutrition counselling to case by nutritionist
- intervention (Experimental): Multi-domain intervention included exercise,cognitive training and diet education was conducted for five hours per week in the first month, second month and third month.
  Interventions: Radiation: health promotion program

INTERVENTIONS:
Radiation: health promotion program — Multi-domain intervention 120 minutes cognitive training, 120 ~180 minutes physical exercise per weeks, and 60 minutes diet nutrition education per month
  Arms: intervention

SUMMARY:
health promotion behavior is important in older adults.The purpose of this study is to examine the efficacy of smart integrated health promotion intervention among middle age adults and older adults in community.

DETAILED DESCRIPTION:
There very limited research focused on leisure activity, nutrition status, quality of life and subjective well-being. In addition, there is lack of research develop smart integrated health promotion intervention to enhance well-being for middle age adults older adults in community and examine the efficacy of the intervention. The purpose of this study is to examine the efficacy of smart integrated health promotion intervention among middle age adults and older adults in community .

ELIGIBILITY:
Inclusion Criteria:

(1) age over 50 years

Exclusion Criteria:

1. those who could not understanding protocol or communication with search nurses;
2. or with cognitive impairment or mental disorders;
3. or advance cancer;
4. or have been myocardial infarction;
5. or congestive heart failure was excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2024-02-17 (Estimated); Study Completion 2024-02-17 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline life quality at 3, 6, 9 month | baseline, 3, 6, 9 month
  measured by the EuroQol- 5 Dimension (EQ-5D), score range 0-1,The higher the score, the better the quality of life
Changes from baseline life quality at 3, 6, 9 month | baseline, 3, 6, 9 month
  measured by the subjective well-being scale, score range 10-50, The higher the score, the better the quality of life

OTHER OUTCOMES:
Changes from baseline one touch blood sugar in mg/dl at 3, 6, 9 month | baseline, 3, 6, 9 month
  Changes from baseline one touch blood sugar in mg/dl at 3, 6, 9 month
Changes from baseline one touch urine acid in mg/dl at 3, 6, 9 month | baseline, 3, 6, 9 month
  Changes from baseline one touch urine acid in mg/dl at 3, 6, 9 month
Changes from baseline one touch total cholesterol in mg/dl at 3, 6, 9 month | baseline, 3, 6, 9 month
  Changes from baseline one touch total cholesterol in mg/dl at 3, 6, 9 month

CONTACTS AND LOCATIONS:
Overall Officials: Heng-Hsin Tung, PhD, Study Director — National Yang Ming Chiao Tung University
Locations (1):
- WISON Pharmacy, Taichung, Taiwan

REFERENCES:
- [Derived] Lee LY, Tung HH, Liao G, Liu SJ, Chen ZY, Yang YR. Multihealth Promotion Programs on Physical Health and Quality of Life in Older Adults: Quasi-Experimental Study. Interact J Med Res. 2025 May 1;14:e65213. doi: 10.2196/65213. PMID 40310677